CLINICAL TRIAL: NCT01038167
Title: An Open-Label Phase 1 Study in Healthy Adult Subjects to Examine the Effects of Telaprevir on the Pharmacokinetics of Cyclosporine and Tacrolimus
Brief Title: A Study to Examine the Effects of Telaprevir on the Pharmacokinetics of Cyclosporine and Tacrolimus in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Robert Kauffman, M.D., Ph.D., Vertex Pharmaceuticals Incorporated
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VX09-950-021
Record Dates: First submitted 2009-12-18; First posted 2009-12-23 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-04

CONDITIONS: Hepatitis C
Keywords: VX-950
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Part A will be administered in two periods, separated by a washout. In Period 1, subjects will receive cyclosporine alone. In Period 2, subjects will receive cyclosporine in combination with telaprevir.
  Interventions: Drug: telaprevir; Drug: cyclosporine
- Part B (Experimental): Part B will be administered in two periods, separated by a washout. In Period 1, subjects will receive tacrolimus alone. In Period 2, subjects will receive tacrolimus in combination with telaprevir.
  Interventions: Drug: telaprevir; Drug: tacrolimus

INTERVENTIONS:
Drug: telaprevir — Tablet, Oral, 750mg, every 8 hours, Day 1-11 of Period 2
  Arms: Part A
Drug: telaprevir — Tablet, Oral, 750mg, every 8 hours, Day 1-13 of Period 2
  Arms: Part B
Drug: cyclosporine — Solution, Oral, 100mg, Day 1 of Period 1
  Arms: Part A
Drug: cyclosporine — Solution, Oral, 10mg, Day 1 and Day 8 of Period 2
  Arms: Part A
Drug: tacrolimus — Capsule, Oral, 2mg, Day 1 of Period 1
  Arms: Part B
Drug: tacrolimus — Capsule, Oral, 0.5mg, Day 8 of Period 2
  Arms: Part B

SUMMARY:
The purpose of this study is to evaluate the effect that telaprevir has on the pharmacokinetics of cyclosporine and tacrolimus. Pharmacokinetics means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female (non-childbearing potential) or male subjects between 18 and 60 years of age (inclusive)
* Body mass index (BMI) from 18 to 30 kg/m2 (inclusive) at the Screening Visit and Day 1, and weigh more than 50 kg at Screening.

Exclusion Criteria:

* History of any illness or condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Participated in a clinical study involving administration of either an investigational or a marketed drug within 2 months or 5 half-lives (whichever is longer) before the Screening Visit.
* Positive result for any of the following infectious disease tests: hepatitis B antigen, hepatitis C virus antibody, human immunodeficiency virus 1 antibody, or human immunodeficiency virus 2 antibody.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Part A only: Pharmacokinetic parameters of cyclosporine (Cmax, AUC0-tlast, AUC0-inf, tmax, t1/2) | 33 days
Part A and Part B: Pharmacokinetic parameters of telaprevir (Cmax, AUC0-8h, Cmin, tmax) | 33 days for Part A; 44 days for Part B
Part B only: Pharmacokinetic parameters of tacrolimus (Cmax, AUC0-tlast, AUC0-inf, tmax, t1/2) | 44 days

SECONDARY OUTCOMES:
Part A and Part B: Safety and tolerability as measured by adverse events, clinical laboratory assessments, electrocardiograms, vital signs, physical examinations | 33 days for Part A; 44 days for Part B

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (1):
- Dallas, Texas, United States